CLINICAL TRIAL: NCT00505908
Title: Non-Interventional F-Two Isoprostane Trial
Brief Title: Non-Interventional F-Two Isoprostane Trial (NIFTI)
Acronym: NIFTI
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Wigginton, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: 052007-034
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Each year in the United States alone, 300,000 persons are hospitalized for traumatic brain injury, with approximately one quarter dying. Despite advances in aggressive neurosurgical interventions, intensive care monitoring and overall supportive management, many of those who do "survive" do not fully recover and are left with a varying degree of permanent disability. It is therefore imperative that new methods of early interventions be explored.

One possible road to effective therapy is to examine the timing of secondary injury via a biological marker, to help guide the timing of treatment directed specifically at early oxidant injury. A more thorough understanding of how quickly oxidant injury occurs will allow us to direct appropriate therapies targeted directly at oxidant injury within what is currently thought to be a very narrow window of opportunity for intervention, possibly peaking within the first two hours after the initial injury.

Potential participants include patients between the ages of 18 and 50 years who are admitted to Parkland Memorial Hospital with a diagnosis of severe traumatic brain injury. Blood, urine, and CSF (if patient requires a clinically indicated ventriculostomy) will be collected over the first 5 days post-injury. Clinically-relevant patient progress, clinically required interventions, neuro-imaging results, and demographics will be tracked while the patient is hospitalized, with final neurological outcome measured at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Estimated age of 18 - 50 years
2. Glasgow Come Scale (GCS) score of between 3 and 8 prior to intubation and/or sedation.
3. Systolic blood pressure of >90 mm Hg
4. Receiving medical treatment in the Emergency Department (ED) of Parkland Hospital, a Level I Trauma Center in Dallas, Texas

Exclusion Criteria:

1. Those in whom the time of injury is unknown
2. Those with any 2 readings of systolic blood pressure of <90 prior to enrollment
3. Those who are known to have legal Do Not Resuscitate (DNR) orders in place prior to enrollment.
4. Those receiving CPR prior to enrollment
5. Known incarcerated individuals
6. Pulse ox reading of < 90 prior to enrollment
7. Status epilepticus prior to enrollment
8. Penetrating head trauma

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who meet inclusion criteria and have experienced a trauamtic head injury.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Levels of oxidant injury in cerebrospinal fluid following severe traumatic brain injury | Up to 5 days
  F2 Isoprostane levels in cerebrospinal fluid following severe traumatic brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Jane G Wigginton, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States